CLINICAL TRIAL: NCT02337634
Title: Silymarin Treatment of Pathological Gambling: A Double-Blind, Placebo-Controlled Study
Brief Title: Milk Thistle in Pathological Gambling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0480
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-02

CONDITIONS: Pathological Gambling; Gambling Disorder
MeSH Terms: conditions — Gambling | interventions — Sugars; milk-thistle extract; Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matched dosage of milk thistle daily.
  Interventions: Drug: Placebo
- Milk Thistle (Active Comparator): Capsule form, 150mg BID to 300mg BID
  Interventions: Drug: Milk Thistle

INTERVENTIONS:
Drug: Placebo — Taken as two 150mg capsules BID for 2 weeks, then 300mg BID for remainder of the study.
  Other Names: Sugar Pill
  Arms: Placebo
Drug: Milk Thistle — Taken as two 150mg capsules BID for 2 weeks, then 300mg BID for remainder of the study.
  Other Names: Silymarin
  Arms: Milk Thistle

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of silymarin in individuals with gambling disorder. The hypothesis to be tested is that silymarin will be more effective and well tolerated in subjects with gambling disorder compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
Gambling disorder is a significant public health problem that often results in a distinctive pattern of persistent and disabling psychological symptoms. Although once thought to be relatively uncommon, studies estimate that gambling disorder has a lifetime prevalence among adults of 1.6% and past-year prevalence of 1.1%. Patients with gambling disorder also experience significant social and occupational impairment as well as financial and legal difficulties.

Individuals with gambling disorder report chronically high levels of stress, and vulnerability to gambling addiction is enhanced by stressful events (4), particularly as stress may result cognitive problems leading to impulsive and unhealthy decisions. A stress response is elicited when sensations and Observations do not match existing or anticipated expectations. A primary endocrine response to stress is the secretion of glucocorticoids through the activation of the hypothalamic-pituitary-adrenal axis. Although their release serves to maintain homeostasis during acute episodes of stress, prolonged stress responses have been associated with structural brain damage both in humans and animals. In humans, stress also enhances addictive craving, and relapse to addiction is more likely to occur in individuals exposed to high levels of stress. Since oxidative stress may be implicated in the etiology of addictive behaviors, use of antioxidants to reduce relapse, improve cognitive functioning, and reduce addictive urges may be a sensible step.

Silymarin, a flavonoid and a member of the Asteraceae family, is extracted from the seeds of milk thistle (Silybum marianum) and is known to own antioxidative and anti-apoptotic properties. Silymarin has been reported to decrease lipid peroxidation. Furthermore, it has been demonstrated that its anti-oxidative activity is related to the scavenging of free radicals and activation of anti-oxidative defenses: increases in cellular glutathione content and superoxide dismutase activity. Milk thistle has been used for a range of psychiatric disorders including methamphetamine abuse and obsessive compulsive disorder, two psychiatric disorders with similarities to gambling disorder. The flavanoid complex silymarin in preclinical studies has been found to increase serotonin levels in the cortex, and ameliorate decreases in dopamine and serotonin in the prefrontal cortex and hippocampus associated with methamphetamine abuse. In the frontal cortex one of the functions of dopamine is to increase the signal to noise ratio, increased dopamine correlating with increased frontal performance. Studies have shown that the higher cortical dopamine levels are associated with improved frontal cortical cognitive performance. Cortical inhibition is felt to be the basis for top-down control of motivated behaviors. A recent randomized controlled study with milk thistle was conducted in Iran Thirty five participants with moderate OCD were randomly assigned to 200 mg of milk thistle leaf extract or 10 mg of fluoxetine three times daily for eight weeks. Results revealed no significant difference in treatment effects between milk thistle and fluoxetine from baseline to endpoint as both interventions provided a highly significant reduction in symptoms.

Silymarin or Milk Thistle may therefore offer promise for the treatment of individuals with gambling disorder. Pharmacological management of gambling symptoms has produced mixed results, with some studies showing a superiority of medication to placebo.

The current pilot study examines the tolerability and efficacy of milk thistle in the treatment of gambling disorder. We hypothesize that milk thistle will reduce the severity of gambling symptoms and improve patients' overall functioning.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-75;
* Diagnosis of current gambling disorder based on DSM-5 criteria and confirmed using the clinician-administered Structured Clinical Interview for Pathological Gambling (SCI-PG) (12);
* Gambling behavior within 2 weeks prior to enrollment;
* Women of child bearing age are required to have a negative result on a beta-human chorionic gonadotropin pregnancy test;
* Women of childbearing potential utilizing a medically accepted form of contraception defined as double barrier, oral contraceptive, injectable contraceptive, implantable contraceptive devices, and abstinence

Exclusion Criteria:

* Infrequent gambling (i.e. less than one time per week) that does not meet DSM-5 criteria for gambling disorder;
* Unstable medical illness or clinically significant abnormalities on laboratory tests, EKG, or physical examination at screen as determined by the investigator;
* History of seizures;
* Myocardial infarction within 6 months;
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
* A need for medication other than milk thistle with possible psychotropic effects or unfavorable interactions as determined by the investigator;
* Clinically significant suicidality (defined by the Columbia Suicidal Scale);
* Lifetime history of bipolar disorder type I or II, schizophrenia, or any psychotic disorder;
* Initiation of psychotherapy or behavior therapy within 3 months prior to study baseline;
* Previous treatment with milk thistle

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Grant JE, Driessens C, Chamberlain SR. Silymarin (Milk Thistle) Treatment of Adults With Gambling Disorder: A Double-Blind, Placebo-Controlled Trial. Clin Neuropharmacol. 2024 Mar-Apr 01;47(2):54-58. doi: 10.1097/WNF.0000000000000585. PMID 38478366
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 enrolled participants were excluded from the study prior to randomization because they did not meet the inclusion criteria.
Period: Overall Study
Arm/Group | Placebo | Milk Thistle
Started | 26 | 17
Completed | 22 | 16
Not Completed | 4 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant assigned to placebo dropped out before being randomized, leaving placebo total at N = 25.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Milk Thistle | Total
Number analyzed (Participants) | 25 | 17 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 16 | 40
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.48 (12.99) | 48.25 (13.64) | 49.6 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 18 | 7 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 4 | 9
  African American | 17 | 13 | 30
  Hispanic/Latino | 1 | 0 | 1
  Native American | 1 | 0 | 1
  Not reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 17 | 42
Yale Brown Obsessive Compulsive Scale Modified for Pathological Gambling (PG-YBOCS) Score [Mean (Standard Deviation); unit: units on a scale] — Every 2 weeks the subject will take the PG-YBOCS for the duration of the 8-week study. At each of these visits the outcome will be assessed, but only one value (change from baseline to week 8) will be reported. The scale itself assess severity of gambling, with higher scores indicating worse outcomes. The scale includes two subscales: a thought/urge subscale and a behavior subscale. Each subscale contains 5 items to be rated with a score of 0-4. Subscale scores are summed to get a total score. Possible total scores range from 0-40.
  units on a scale | 20.62 (3.40) | 21.17 (3.1) | 20.84 (3.36)

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Pathological Gambling (PG-YBOCS)
Description: Every 2 weeks the subject will take the PG-YBOCS for the duration of the 8-week study. At each of these visits the outcome will be assessed, but only one value (change from baseline to week 8) will be reported. The scale itself assesses severity of gambling, with higher scores indicating worse outcomes. The scale includes two subscales: a thought/urge subscale and a behavior subscale. Each subscale contains 5 items to be rated with a score of 0-4. Subscale scores are summed to get a total score. Possible total scores range from 0-40.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had PG-YBOCS data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 21 | 16
units on a scale | -11.76 (7.18) | -11.86 (7.75)

2. Secondary Outcome: Clinical Global Impression-Improvement and Severity Scales (CGI-I and CGI-S)
Description: The entire study for an individual subject will last 8 weeks. Every 2 weeks the subject will take the CGIs for the duration of the 8 weeks. Results are reported as the change in Week 8-Week 0 scores. The scales themselves assess overall disorder severity, with higher scores indicating worse outcomes (i.e., less improvement or greater severity). Possible total scores range from 1-7.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: There was less participant data analyzed for the CGI-S because several participants were missing this data either for their first or last study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 21 | 14
units on a scale
  Change in CGI-I score | -0.90 (1.67) | -1.71 (1.14)
  Change in CGI-S score: number analyzed (Participants) | 8 | 6
  Change in CGI-S score | -1.5 (1.41) | -1.5 (1.38)

3. Secondary Outcome: Gambling Symptom Assessment Scale (G-SAS)
Description: Every 2 weeks the subject will take the G-SAS for the duration of the 8-week study. This is a 12-item, reliable and valid, self-rated scale assessing gambling urges, thoughts, and behaviors during the previous seven days. At each of these visits the outcome will be assessed, but only one value (change from baseline to week 8) will be reported. The scale itself assess severity of gambling symptoms, with a higher score indicating a worse outcome. Each item can be rated with a score of 0-4, with the sum of the 12 items equaling the total score. Possible total scores range from 0-48.
Time Frame: Once every two weeks for the 8 weeks of the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 22 | 15
units on a scale | -15.54 (9.91) | -19.72 (8.55)

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The entire study for an individual subject will last 8 weeks. Every 2 weeks the subject will take the HAM-A for the duration of the 8 weeks. Results are reported as the change in Week 8-Week 0 scores. The scale itself assess levels of anxiety, with higher scores indicating worse outcomes. Possible total scores range from 0-56.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had HAM-A data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 9 | 7
units on a scale | -3 (2.5) | -0.43 (0.96)

5. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The entire study for an individual subject will last 8 weeks. Every 2 weeks the subject will take the SDS for the duration of the 8 weeks. Results are reported as the change in Week 8-Week 0 scores. The scale itself assesses level of disability resulting from gambling (or target disorder), with higher scores indicating worse outcomes. Possible total scores range from 0-30.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had SDS data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 17 | 13
units on a scale | -9.94 (10.15) | -8 (9.57)

6. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The entire study for an individual subject will last 8 weeks. Every 2 weeks the subject will take the HAM-D for the duration of the 8 weeks. Results are reported as the change in Week 8-Week 0 scores. The scale itself assesses level of depression, with higher scores indicating worse outcomes. Possible total scores range from 0-52.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had HAM-D data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 9 | 6
units on a scale | -2.56 (2.51) | -2.33 (2.07)

7. Secondary Outcome: Perceived Stress Scale (PSS)
Description: The entire study for an individual subject will last 8 weeks. Every 2 weeks the subject will take the PSS for the duration of the 8 weeks. Results are reported as the change in Week 8-Week 0 scores. The scale itself assesses the level of perceived stress the individual experiences, with higher scores indicating worse outcomes. Possible total scores range from 0-40.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had PSS data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 9 | 8
units on a scale | -5.44 (3.84) | -3.88 (5.99)

8. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: The entire study for an individual subject will last 8 weeks. This inventory will be completed at the first and last visit of the study, with only these two points being assessed. Results are reported as the change in Week 8-Week 0 scores. The scale itself assess the subjects overall perceived quality of life, with higher scores indicating better outcomes. Possible total scores range from 1-77.
Time Frame: Once every two weeks for the 8 weeks of the study
Population: Participants who had QOLI data at Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Milk Thistle
Number analyzed (Participants) | 13 | 10
units on a scale | 10.92 (28.61) | 1.3 (41.42)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time participants signed consent until their final Week 8 visit.
Description: The definition of adverse events in this study matches the clinicaltrials.gov definition.
Arm/Group | Placebo | Milk Thistle
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/17
Other Adverse Events (participants affected / at risk) | 3/26 | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Milk Thistle (N=17)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reduced appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 0 (0)
Increased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limited statistical power due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02337634/Prot_SAP_000.pdf